CLINICAL TRIAL: NCT00971672
Title: Incidence of Iron Deficiency Anemia in Toddlers
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Dr Koren Ariel, Head of Pediatric Hematology Unit and Pediatric Dpt B, HaEmek Medical Center, Israel
Other Study IDs: 0024/09-EMC
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Healthy Infants
Keywords: Infants; Iron Deficiency; Anemia; Healthy infants that attend the pediatric community clinics
MeSH Terms: conditions — Iron Deficiencies; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Toddlers from Jewish origin: Toddlers from Jewish origin aged 18 to 36 months
  Interventions: Other: Questionnaire filling and laboratory analysis
- Toddlers from non Jewish origin: Toddlers aged 18 to 36 months belonging to non Jewish (Arab) population
  Interventions: Other: Questionnaire filling and laboratory analysis

INTERVENTIONS:
Other: Questionnaire filling and laboratory analysis — A questionnaire that included demographic characteristics, nutrition and iron supplementation in the first year, growth status, and laboratory results will be filled for each patient.
  The laboratory analysis will include complete blood count and serum ferritin analysis.

SUMMARY:
The frequency of iron deficiency anemia was extensively studied in infants on the first year of life. There is not enough information about the frequency of iron deficiency during the second and third years of life. In a previous study performed in Israel and published in Pediatrics 2006 the incidence of anemia does not decrease towards age 18 months. Then there is reasonable to study the iron deficiency frequency beyond this age.

DETAILED DESCRIPTION:
The purpose of this study is to analyze the frequency of Iron deficiency anemia in a group of 400 toddles from age 18 months to 36 months.

Two groups of children will be included, 200 children from Jewish origin and 200 from non Jewish origin, mostly Arabs.

A questionnaire that included demographic characteristics, nutrition and iron supplementation in the first year, growth status, and laboratory results will be filled for each patient.

The laboratory analysis will include complete blood count and serum ferritin analysis.

Children that were previously diagnosed suffering from iron deficiency, children suffering from chronic diseases or were born premature will not be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children that attend the pediatric community clinics.

Exclusion Criteria:

* Children that were previously diagnosed suffering from iron deficiency.
* Children suffering from chronic diseases or were born premature will not be included in the study.

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The purpose of this study is to analyze the frequency of Iron deficiency anemia in a group of 400 toddles from age 18 months to 36 months.
  Two groups of children will be included, 200 children from Jewish origin and 200 from non Jewish origin, mostly Arabs.
  Children that were previously diagnosed suffering from iron deficiency, children suffering from chronic diseases or were born premature will not be included in the study.
Sampling Method: Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2010-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Frequency of anemia (Hemoglobin below normal for age) and Iron deficiency (Low ferritin value) | One year

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Koren, MD, Principal Investigator — Pediatric Dpt B and Pediatric Hemaology Unit - Ha'Emek Medical Center - Afula - Israel
Locations (1):
- Pediatric Hematology Unit - Ha'Emek Medical Center, Afula, Afula, Israel